CLINICAL TRIAL: NCT05050968
Title: Effects of Controlled Physical Activity on the Fitness, Body Composition and Quality of Life of Obese Women Undergoing Bariatric Surgery
Brief Title: Physical Activity and Bariatric Surgery
Acronym: ACTIBARIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHRO-2016-03
Record Dates: First submitted 2021-07-22; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Bariatric Surgery Candidate
Keywords: Physical activity; Bariatric Surgery; Physical Fitness; Quality of life; Body Composition
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study is an open-label, randomized, single-center trial with two groups: an Adapted Physical Activity group and a control group performing no controlled physical activity within each group women undergoing bypass or sleeve surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity Group (Experimental): Patients will follow a 3-month physical activity program 3 times a week between V1 and V2. Then, between V2 and V3, no APA program will be offered to both groups.
  Interventions: Other: Physical activity
- Control group (No Intervention): Patients will receive standard hospital management

INTERVENTIONS:
Other: Physical activity — Between V1 and V2 (i.e. 12 weeks), the APAG (Adapted Physical Activity Group) will participate at a physical training program, 3 sessions of 1h30 per week consisting of endurance activities (60-75% of VO2 peak) and muscle strengthening while the CG will not perform any controlled physical training program. Then, between V2 and V3, no APA (Adapted Physical Activity) program will be offered to both groups.
  Arms: Adapted Physical Activity Group

SUMMARY:
Bariatric surgery indeed leads to significant weight loss, reduces mortality risk, obesity-associated comorbidities (Wolfe et al., 2016) and improves functional physical abilities (Herring et al., 2016). Because these benefits are related to decreased energy intake, the investigators aim to optimize them by combining them with supervised adapted physical activity practice.

So, the aim of this clinical trial is to measure the effects of a physical training program on physical fitness, body composition and quality of life of obese women who have undergone bariatric surgery.

DETAILED DESCRIPTION:
Upon hospitalization for their bariatric surgery (bypass or sleeve), subjects will sign their informed consent and be included in the study. Six weeks' post-surgery, the subjects will be randomized in one of the 2 groups (Control group CG or Adapted Physical Activity group APAG). Patients in both groups will have 3 postoperative visits one at 6 weeks (V1), one at 18 weeks (V2) and one at 30 weeks (V3). During these visits, they will undergo the same assessments (body composition, physical condition, quality of life). Patients in the CG will receive standard hospital management. Patients in APAG will follow the same management and will also follow a 3-month physical activity program 3 times a week between V1 and V2. Then, between V2 and V3, no APA program will be offered to both groups.

The subjects will evaluate during each visit V1, V2 and V3:

* body composition,
* physical condition,
* quality of life
* daily physical activity

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 55 years old
* undergoing bariatric surgery (a "bypass gastric" or a "sleeve")
* not practicing a supervised physical activity
* having read and signed an informed consent prior to the start of the trial
* being affiliated to a social security system

Exclusion Criteria:

* Women with a contraindication to physical activity
* any medical contraindication to the practice of stress tests.
* unable to go to the hospital regularly
* having a significant functional limitation that does not allow her to perform the 6-minute walk test
* with an intellectual disability and/or psychiatric illness
* does not speak and/or understand French
* pregnant woman
* under guardianship or curatorship
* participating in another clinical research

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen consumption (VO2 max) | Week 6
  The VO2 max is measured during an effort test with progressively increasing and maximum load which consists in making the subject pedal against an increasing load
Maximum oxygen consumption (VO2 max) | Week 18
  The VO2 max is measured during an effort test with progressively increasing and maximum load which consists in making the subject pedal against an increasing load
Maximum oxygen consumption (VO2 max) | Week 30
  The VO2 max is measured during an effort test with progressively increasing and maximum load which consists in making the subject pedal against an increasing load

SECONDARY OUTCOMES:
Impact of obesity on the physical, psycho-social, dietary well-being and dieting experience assessed using the Quality of Life, Obesity and Diet Scale (QOLDS) | Week 6
  QoL will be assessed using a simplified version of the French obesity-specific QoL questionnaire developed by Ziegler et al. Each participant will be asked to evaluate 14 statements about their life on a 4-point Likert scale (with 1 representing total disagreement and 4 representing total agreement). The 14 statements (eg, "Because of my weight, I have trouble to dress or undress") will equally be divided between physical aspects of life and psychosocial aspects of life. A French obesity-specific QoL questionnaire will be used to calculate the participants' physical dimension of QoL scores and psychoso-cial dimension of QoL scores by summing the points for each relevant item (range: 7-28 points). The total score will also be calculated (range: 14-56 points). The higher the scores, the better the QoL.
Impact of obesity on the physical, psycho-social, dietary well-being and dieting experience assessed using the Quality of Life, Obesity and Diet Scale (QOLDS) | Week 18
  QoL will be assessed using a simplified version of the French obesity-specific QoL questionnaire developed by Ziegler et al. Each participant will be asked to evaluate 14 statements about their life on a 4-point Likert scale (with 1 representing total disagreement and 4 representing total agreement). The 14 statements (eg, "Because of my weight, I have trouble to dress or undress") will equally be divided between physical aspects of life and psychosocial aspects of life. A French obesity-specific QoL questionnaire will be used to calculate the participants' physical dimension of QoL scores and psychoso-cial dimension of QoL scores by summing the points for each relevant item (range: 7-28 points). The total score will also be calculated (range: 14-56 points). The higher the scores, the better the QoL.
Impact of obesity on the physical, psycho-social, dietary well-being and dieting experience assessed using the Quality of Life, Obesity and Diet Scale (QOLDS) | Week 30
  QoL will be assessed using a simplified version of the French obesity-specific QoL questionnaire developed by Ziegler et al. Each participant will be asked to evaluate 14 statements about their life on a 4-point Likert scale (with 1 representing total disagreement and 4 representing total agreement). The 14 statements (eg, "Because of my weight, I have trouble to dress or undress") will equally be divided between physical aspects of life and psychosocial aspects of life. A French obesity-specific QoL questionnaire will be used to calculate the participants' physical dimension of QoL scores and psychoso-cial dimension of QoL scores by summing the points for each relevant item (range: 7-28 points). The total score will also be calculated (range: 14-56 points). The higher the scores, the better the QoL.
Walking distance | Week 6
  The walking distance (meters) will be evaluated during the 6 minutes walk test
Walking distance | Week 18
  The walking distance (meters) will be evaluated during the 6 minutes walk test
Walking distance | Week 30
  The walking distance (meters) will be evaluated during the 6 minutes walk test
Heart rate | Week 6
  The heart rate (beats/min) will be evaluated during the 6 minutes walk test
Heart rate | Week 18
  The heart rate (beats/min) will be evaluated during the 6 minutes walk test
Heart rate | Week 30
  The heart rate (beats/min) will be evaluated during the 6 minutes walk test
Perception of the effort | Week 6
  This will be evaluated with a Borg scale (the minimum score is 0 = no exertion and the maximal 10 = maximal exertion) at the end of the 6-minutes walk test.
Perception of the effort | Week 18
  This will be evaluated with a Borg scale (the minimum score is 0 = no exertion and the maximal 10 = maximal exertion) at the end of the 6-minutes walk test.
Perception of the effort | Week 36
  This will be evaluated with a Borg scale (the minimum score is 0 = no exertion and the maximal 10 = maximal exertion) at the end of the 6-minutes walk test.
Maximum voluntary force of the quadriceps | week 6
  The maximum voluntary isometric strength of the knee extensors (strength of quadriceps in kilograms) will be measured with a MicroFET2 handheld dynamometer.
  Each participant's lower extremity could be placed in a position a knee flexion of 90 degrees. They will be asked to apply maximal force against the dynamometer held by the physical therapist. Before the test, the participants will be given a standard instruction of "push as hard as you can." Encouragement to apply maximal effort will also be given during the test. Each participant will be instructed to exert maximal strength for 3-5 seconds until the examiner instructed the patient to relax.
Maximum voluntary force of the quadriceps | week 18
  The maximum voluntary isometric strength of the knee extensors (strength of quadriceps in kilograms) will be measured with a MicroFET2 handheld dynamometer.
  Each participant's lower extremity could be placed in a position a knee flexion of 90 degrees. They will be asked to apply maximal force against the dynamometer held by the physical therapist. Before the test, the participants will be given a standard instruction of "push as hard as you can." Encouragement to apply maximal effort will also be given during the test. Each participant will be instructed to exert maximal strength for 3-5 seconds until the examiner instructed the patient to relax.
Maximum voluntary force of the quadriceps | week 30
  The maximum voluntary isometric strength of the knee extensors (strength of quadriceps in kilograms) will be measured with a MicroFET2 handheld dynamometer.
  Each participant's lower extremity could be placed in a position a knee flexion of 90 degrees. They will be asked to apply maximal force against the dynamometer held by the physical therapist. Before the test, the participants will be given a standard instruction of "push as hard as you can." Encouragement to apply maximal effort will also be given during the test. Each participant will be instructed to exert maximal strength for 3-5 seconds until the examiner instructed the patient to relax.
grip strength | week 6
  The grip strength will be evaluated with a dynamometer that can be squeezed very hard for 3 seconds. The measurement will be evaluated three times with 30 seconds of recovery and the maximum value will be retained.
grip strength | week 18
  The grip strength will be evaluated with a dynamometer that can be squeezed very hard for 3 seconds. The measurement will be evaluated three times with 30 seconds of recovery and the maximum value will be retained.
grip strength | week 30
  The grip strength will be evaluated with a dynamometer that can be squeezed very hard for 3 seconds. The measurement will be evaluated three times with 30 seconds of recovery and the maximum value will be retained.
Body composition | week 6
  Body composition will be assessed by a body composition analyser in the morning on an empty stomach
Body composition | week 18
  Body composition will be assessed by a body composition analyser in the morning on an empty stomach
Body composition | week 30
  Body composition will be assessed by a body composition analyser in the morning on an empty stomach
Metabolic measurements | week 6
  During the constant workload exercise, blood samples will be taken and metabolic measurements will be made:
  - Blood Lactate (mmol/L)
Metabolic measurements | week 6
  During the constant workload exercise, blood samples will be taken and metabolic measurements will be made:
  - Blood glucose (g/L)
Hormonal measurements | week 6
  During the constant workload exercise, blood samples will be taken and hormonal measurements will be made:
  * Testosterone (ng/ml)
  * Cortisol (ng/ml)
Metabolic measurements | week 18
  During the constant workload exercise, blood samples will be taken and metabolic measurements will be made:
  - Blood glucose (g/L)
Metabolic measurements | week 18
  During the constant workload exercise, blood samples will be taken and metabolic measurements will be made:
  - Blood Lactate (mmol/L)
Hormonal measurements | week 18
  During the constant workload exercise, blood samples will be taken and hormonal measurements will be made:
  * Testosterone (ng/ml)
  * Cortisol (ng/ml)
Metabolic measurements | week 30
  During the constant workload exercise, blood samples will be taken and metabolic measurements will be made:
  - Blood glucose (g/L)
Metabolic measurements | week 30
  During the constant workload exercise, blood samples will be taken and metabolic measurements will be made:
  - Blood Lactate (mmol/L)
Hormonal measurements | week 30
  During the constant workload exercise, blood samples will be taken and hormonal measurements will be made:
  * Testosterone (ng/ml)
  * Cortisol (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Virgile AMIOT, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Baillot A, Audet M, Baillargeon JP, Dionne IJ, Valiquette L, Rosa-Fortin MM, Abou Chakra CN, Comeau E, Langlois MF. Impact of physical activity and fitness in class II and III obese individuals: a systematic review. Obes Rev. 2014 Sep;15(9):721-39. doi: 10.1111/obr.12171. Epub 2014 Apr 9. PMID 24712685
- [Background] Berggren JR, Boyle KE, Chapman WH, Houmard JA. Skeletal muscle lipid oxidation and obesity: influence of weight loss and exercise. Am J Physiol Endocrinol Metab. 2008 Apr;294(4):E726-32. doi: 10.1152/ajpendo.00354.2007. Epub 2008 Feb 5. PMID 18252891
- [Background] Blair SN, Cheng Y, Holder JS. Is physical activity or physical fitness more important in defining health benefits? Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S379-99; discussion S419-20. doi: 10.1097/00005768-200106001-00007. PMID 11427763
- [Background] Bond DS, Phelan S, Wolfe LG, Evans RK, Meador JG, Kellum JM, Maher JW, Wing RR. Becoming physically active after bariatric surgery is associated with improved weight loss and health-related quality of life. Obesity (Silver Spring). 2009 Jan;17(1):78-83. doi: 10.1038/oby.2008.501. Epub 2008 Nov 6. PMID 18997679
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Wolfe BM, Kvach E, Eckel RH. Treatment of Obesity: Weight Loss and Bariatric Surgery. Circ Res. 2016 May 27;118(11):1844-55. doi: 10.1161/CIRCRESAHA.116.307591. PMID 27230645
- [Background] Herring LY, Stevinson C, Davies MJ, Biddle SJ, Sutton C, Bowrey D, Carter P. Changes in physical activity behaviour and physical function after bariatric surgery: a systematic review and meta-analysis. Obes Rev. 2016 Mar;17(3):250-61. doi: 10.1111/obr.12361. Epub 2016 Jan 18. PMID 26783103